CLINICAL TRIAL: NCT03590574
Title: A Single Arm, Open Label, Multi-centre, Phase I/II Study Evaluating the Safety and Clinical Activity of AUTO4, a CAR T-cell Treatment Targeting TRBC1, in Patients With Relapsed or Refractory TRBC1 Positive Selected T Cell Non-Hodgkin Lymphoma
Brief Title: Phase I/II Study Evaluating AUTO4 in Patients With TRBC1 Positive T Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Autolus Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTO4-TL1; 2017-001965-26 (EudraCT Number)
Record Dates: First submitted 2018-07-07; First posted 2018-07-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: T Cell Non-Hodgkin Lymphoma; Peripheral T-Cell Lymphoma, Not Otherwise Specified; Angioimmunoblastic T-cell Lymphoma; Anaplastic Large Cell Lymphoma
Keywords: T cell lymphoma; Relapsed T cell Non-Hodgkin Lymphoma; Refractory T cell Non-Hodgkin Lymphoma; AUTO4
MeSH Terms: conditions — Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AUTO4 (Experimental): Relapsed or refractory T cell non-Hodgkin Lymphoma patients
  Interventions: Biological: AUTO4

INTERVENTIONS:
Biological: AUTO4 — AUTO4 (RQR8/aTRBC1 CAR T cells) Following pre-conditioning with chemotherapy (cyclophosphamide and fludarabine), patients will be treated with doses from 25 to 900 x 10^6 RQR8/aTRBC1 CAR T cells in Phase I. Following dose determination patients will be treated with the selected doses of RQR8/aTRBC1 CAR T cells (AUTO4) in Phase II.

SUMMARY:
The purpose of this study is to test the safety and efficacy of AUTO4 a CAR T cell treatment targeting TRBC1 in patients with relapsed or refractory TRBC1 positive selected T-Non-Hodgkin Lymphoma.

DETAILED DESCRIPTION:
The study will consist of 2 phases, a Phase I/dose escalation phase and a Phase II/expansion phase. Patients with relapsed or refractory TRBC1 positive selected T-NHL will be enrolled in both phases of the study. Eligible patients will undergo leukapheresis to harvest T cells, the starting material for the manufacture of the autologous CAR-T product AUTO4. Following preconditioning by a chemotherapeutic regimen, the patient will receive AUTO4 intravenously as a single dose following which they will then enter a 24-month follow-up period

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years.
2. Willing and able to give written, informed consent to be screened for TRBC1 positive T-NHL and to enter the main study.
3. Confirmed diagnosis of selected T-NHL, including:

   1. Peripheral T cell lymphoma NOS, or
   2. Angioimmunoblastic T cell lymphoma, or
   3. Anaplastic large cell lymphoma
4. Confirmed TRBC1 positive tumour.
5. Relapsed or refractory disease and have had ≥1 prior lines of therapy.
6. Positron emission tomography (PET)-positive measurable disease per Lugano classification.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
8. Adequate bone marrow function without the requirement for ongoing blood products and meets the following criteria:

   1. Absolute neutrophil count ≥1.0 x 109/L
   2. Absolute lymphocyte count ≥0.5 x 109/L (at entry and prior to leukapheresis).
   3. Haemoglobin ≥80 g/L
   4. Platelets ≥75 x 109/L
9. Adequate renal, hepatic, pulmonary, and cardiac function defined as:

   1. Creatinine clearance (as estimated by Cockcroft Gault) ≥60 cc/min.
   2. Serum alanine aminotransferase/aspartate aminotransferase ≤2.5 x upper limit of normal (ULN).
   3. Total bilirubin ≤25 µmol/L (1.5 mg/dL), except in patients with Gilbert's syndrome.
   4. Left ventricular ejection fraction (LVEF) ≥50% by echocardiogram (ECHO) or multiple gated acquisition (MUGA) cardiac scan, unless the institutional lower limit of normal is lower.
   5. Baseline oxygen saturation ≥92% on room air and ≤Grade 1 dyspnoea.
10. For females of childbearing potential (defined as <2 years after last menstruation or not surgically sterile), a negative serum or urine pregnancy test must be documented at screening, prior to pre-conditioning and confirmed before receiving the first dose of study treatment. For females who are not postmenopausal (<24 months of amenorrhea) or who are not surgically sterile (absence of ovaries and/or uterus), a highly effective method of contraception together with a barrier method must be used from the start of the pre-conditioning stage and for at least 12 months after the last dose of AUTO4 (study treatment). They must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 12 months after receiving the last dose of study drug
11. For males, it must be agreed that two acceptable methods of contraception are used.
12. No contra-indications for leukapheresis, or the pre-conditioning regimen.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria must not be enrolled into the study:

1. Patients with T cell leukaemia.
2. Females who are pregnant or lactating.
3. Prior treatment with investigational gene therapy or approved gene therapy or genetically engineered cell therapy product or allogeneic stem cell transplant.
4. Known history or presence of clinically relevant central nervous system (CNS) pathology. Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the CNS.
5. Current or history of CNS involvement by malignancy.
6. Clinically significant, uncontrolled heart disease

   1. Uncontrolled cardiac arrhythmia (patients with rate-controlled atrial fibrillation are not excluded).
   2. Evidence of pericardial effusion.
7. Patients with evidence of uncontrolled hypertension or with a history of hypertension crisis or hypertensive encephalopathy.
8. Patients with a history (within 3 months) or evidence of deep vein thrombosis or pulmonary embolism requiring ongoing therapeutic anticoagulation at the time of pre-conditioning.
9. Patients with active gastrointestinal (GI) bleeding.
10. Patients with any major surgical intervention in the last 3 months.
11. Active infectious bacterial, viral disease or fungal disease (hepatitis B virus, hepatitis C virus, human immunodeficiency virus [HIV], human T cell lymphotropic virus [HTLV] or syphilis) requiring treatment.
12. Active autoimmune disease requiring immunosuppression.
13. History of other neoplasms unless disease free for at least 2 years (adequately treated carcinoma in situ, curatively treated non-melanoma skin cancer, breast or prostate cancer on hormonal therapy are allowed).
14. Prior treatment with programmed cell death protein 1 (PD1), programmed death ligand 1 (PD-L1), or cytotoxic T lymphocyte-associated protein 4 (CTLA-4) targeted therapy, or tumour necrosis factor (TNF) receptor superfamily agonists including CD134 (OX40), CD27, CD137 (41BB), and CD357 (glucocorticoid induced TNF receptor family related protein) within 6 weeks prior to AUTO4 infusion.
15. The following medications are excluded:

    1. Steroids: Therapeutic doses of prednisone/equivalent of more than 20 mg per day are prohibited within 7 days prior to leukapheresis or pre-conditioning chemotherapy administration. However, physiological replacement, topical and inhaled steroids are permitted.
    2. Cytotoxic chemotherapies within 2 weeks prior to leukapheresis or AUTO4 infusion.
    3. Antibody therapy use within 2 weeks prior to AUTO4 infusion, or five half-lives of the respective antibody, whichever is shorter.
    4. Live vaccine within 4 weeks prior to enrolment.
16. Research participants receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy.
17. Use of rituximab (or rituximab biosimilar) within the last 6 months prior to AUTO4 infusion.
18. Patients, who in the opinion of the Investigator, may not be able to understand or comply with the safety monitoring requirements of the study.

For pre-conditioning chemotherapy and AUTO4 Infusion: Patients meeting any of the following exclusion criteria must not be treated with pre-conditioning chemotherapy or

AUTO4 - and have treatment delayed until they no longer meet these criteria:

1. Severe intercurrent infection at the time of pre-conditioning chemotherapy or the scheduled AUTO4 infusion.
2. Requirement for supplementary oxygen or active pulmonary infiltrates or significant deterioration of organ function at the time of pre-conditioning chemotherapy or scheduled AUTO4 infusion.
3. Significant clinical deterioration of organ functions from screening, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Phase I: Safety (Frequency and severity of adverse events and serious AEs) and confirmation of Phase II dose and schedule. | 24 months post treatment
Phase II: Objective Response (CR + PR) Rate post AUTO4 infusion. | 24 months post treatment

SECONDARY OUTCOMES:
Assess overall safety and tolerability in terms of frequency and severity of all AEs and SAEs and incidence and severity of opportunistic infections following AUTO4 infusion. | 24 months post treatment
Feasibility of generating AUTO4: Number of patients whose cells achieve successful AUTO4 manufacture as a proportion of the number of patients undergoing leukapheresis. | Up to 8 weeks post leukapheresis
Time to response (PR and CR) | 24 months post treatment

CONTACTS AND LOCATIONS:
Locations (5):
- Vall d'Hebron Institute of Oncology, Barcelona, Spain
- United Kingdom (4):
  - Queen Elizabeth University Hospital, Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - Manchester Royal Infirmary Hospital, Manchester
  - Freeman Hospital, The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cwynarski K, Iacoboni G, Tholouli E, Menne T, Irvine DA, Balasubramaniam N, Wood L, Shang J, Xue E, Zhang Y, Basilico S, Neves M, Raymond M, Scott I, El-Kholy M, Jha R, Dainton-Smith H, Hussain R, Day W, Ferrari M, Thomas S, Lilova K, Brugger W, Marafioti T, Lao-Sirieix P, Maciocia P, Pule M. TRBC1-CAR T cell therapy in peripheral T cell lymphoma: a phase 1/2 trial. Nat Med. 2025 Jan;31(1):137-143. doi: 10.1038/s41591-024-03326-7. Epub 2024 Nov 11. PMID 39528665